CLINICAL TRIAL: NCT03668093
Title: Evaluation of CAMBRA Versus ICCMS Caries Risk Assessment Models Acquisition On Treatment Plan In Young Adult Population
Brief Title: Evaluation of CAMBRA Versus ICCMS Caries Risk Assessment Models Acquisition On Treatment Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yomna sayed khallaf, demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-07
Record Dates: First submitted 2018-09-08; First posted 2018-09-12 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Dental Caries
Keywords: caries prevention; caries management
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICCMS (Experimental): Intervention
  Interventions: Other: CAMBRA
- CAMBRA (Active Comparator): Comparator
  Interventions: Other: ICCM

INTERVENTIONS:
Other: ICCM — comprehensive system for caries management
  Arms: CAMBRA
Other: CAMBRA — Caries risk assessment model
  Arms: ICCMS

SUMMARY:
randomized clinical study to evaluate 'caries management by risk assessment' Versus 'international caries classification and management system' Caries Risk Assessment Models Acquisition On Treatment Plan In Young Adult Population with null hypothesis that International Caries Classification and Management System (ICCMS™) will have the same clinical performance as Caries management by risk assessment (CAMBRA)

DETAILED DESCRIPTION:
. (ICCMS™) Comprehensive Patient Care Pathway considered as significant development from the traditional system of treatment plan. Comprehensive patient care should include all recent information related to the biological, social, behavioral, cultural, systemic, and dental/oral risk factors which help development and progression of dental caries. (ICCMS™) also report all essential decisions that aid to preserve tooth structure; as diagnosis, prevention and restoration only if indicated [9]. Moreover ( ICCMS™) deals with caries as a disease and not as a lesion, prevent development of initial caries lesions, and restore moderate or extensive caries lesions with the aim of preserving of tooth structure as much as possible.

Follow up period is selected to be 12 months, since risk category is changed for better or worse over 1-2 year.

ELIGIBILITY:
Inclusion Criteria:

* New patients
* Able to give informed consent in Arabic
* Unlikely to move from the area within 1y for work educational, or personal reasons (determined by residential history and questioning);
* Willing to participate regardless of group assignment
* Willing to comply with all study procedures and protocol
* ≥16 permanent teeth

Exclusion Criteria:

* Patient not willing to have dental radiographs taken
* Patient with significant past or current medical conditions that might affect oral health or oral flora (i.e., diabetes, human immunodeficiency virus, heart conditions requiring antibiotic prophylaxis)
* Patient with medication use that might affect the oral flora or salivary flow (e.g., antibiotic use in the past 3 months, drugs associated with dry mouth/xerostomia)
* Patient with root caries at enrollment
* Patient with periodontal disease requiring surgery, chemotherapeutic agents, or frequent prophylaxis

Ages: 17 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
new carious lesions | 12 months
  Primary outcome :-New carious lesions Measuring device:- Visual-Tactile & Digital radiograph "Digora" Measuring unit :- Scoring system (ordinal)
  (ICDASTM code 0) Sound surfaces
  Initial stage caries (ICDASTM codes 1 and 2) First or distinct visual changes in enamel seen as a carious opacity or visible discolouration Moderate stage caries (ICDASTM codes 3 and 4) A white or brown spot lesion with Localised enamel breakdown, without visible dentine exposure (ICDASTM code 3), or an Underlying dentine shadow (ICDASTM code 4) Extensive stage caries (ICDASTM codes 5 and 6) A distinct cavity in opaque or discoloured enamel with visible dentine (ICDASTM code 5 or 6).

CONTACTS AND LOCATIONS:
Overall Officials: Yomna Khallaf, MD, Principal Investigator — Cairo University
Locations (1):
- Yomna, Cairo, Egypt